CLINICAL TRIAL: NCT04402918
Title: Study of Viral Load and Maternal-fetal Serology in the Interpretation of the Vertical Transmission of SARS Cov-2 During Pregnancy
Brief Title: Study of Viral Load and Maternal-fetal Serology in the Interpretation of the Vertical Transmission of SARS Cov-2 (COVID-19) During Pregnancy
Acronym: TRANSCOVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020/500
Record Dates: First submitted 2020-05-18; First posted 2020-05-27 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Sars-CoV2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pregnancy patients diagnosed with SARS Cov2 during pregnancy (Other): Delivery day biological samples from the mother and the newborn will be performed
  Interventions: Diagnostic Test: biological samples day of delivery

INTERVENTIONS:
Diagnostic Test: biological samples day of delivery — mother samples: serology, viremia, nasopharyngeal swab, vaginal swab, placenta swab, piece of placenta newborn: serology, viremia, nasopharyngeal aspiration

SUMMARY:
The study evaluates the distribution of immunological and virological profiles of newborns patients. Mothers of these children have a proven infection to SARS Cov-2 during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* pregnant woman
* diagnosed with Sars Cov-2 during pregnancy
* singleton or twin pregnancy
* informed consent

Exclusion Criteria:

* virological or serological samples not done the day of delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women
Enrollment: 160 (Actual)
Dates: Start 2020-05-17 (Actual); Primary Completion 2020-05-19 (Actual); Study Completion 2021-08-02 (Actual)

PRIMARY OUTCOMES:
Vrological profile of newborns. | day of delivery
  Describe the virological profile of newborns whose mother have been diagnosed with Sars Cov2 during pregnancy : Covid+ or covid-
Immunological profile of newborns. | day of delivery
  Describe the immunological profile of newborns whose mother have been diagnosed with Sars Cov2 during pregnancy : IgG and/or IgM or absence

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Besancon, Besançon, France

IPD SHARING:
Plan to Share IPD: No